CLINICAL TRIAL: NCT00834652
Title: Improving Depression Treatment Outcomes With an Insulin-Sensitizing Agent
Brief Title: Adding an Insulin-Sensitizing Medication to Depression Treatment for People Who Are Depressed and Overweight
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH081150 (NIH); R01MH081150 (NIH); DAHBR 96-BHC
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Depression
Keywords: Metabolic Diseases; Depressive Disorder, Major; Depressive Disorder; Glucose Metabolism Disorders; Depression Recurrence
MeSH Terms: conditions — Depression; Metabolic Diseases; Depressive Disorder, Major; Depressive Disorder; Glucose Metabolism Disorders | interventions — Sertraline; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive sertraline and metformin.
  Interventions: Drug: Sertraline; Drug: Metformin
- 2 (Placebo Comparator): Participants will receive sertraline and placebo.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — 50 mg once a day, which may be increased to 200 mg once a day
  Other Names: Zoloft
Drug: Metformin — Starting dose of 500 mg daily and increasing by 500 mg every 2 weeks to a total of 2,000 mg daily
  Arms: 1

SUMMARY:
This study will determine whether the drug metformin improves the effects of traditional antidepressant medications in people who are overweight.

DETAILED DESCRIPTION:
Current depression treatments are not effective for approximately one-half of overweight people, and depression eventually returns in approximately one-third of those overweight people whose initial treatment is effective. One possible reason for these treatment failures is that overweight people often experience a condition called insulin resistance (IR), which can lead to type 2 diabetes, an associated disease that might also affect depression treatment. IR results in elevated blood sugar levels that may interfere with medications used to treat depression. Metformin, a medication commonly used to treat diabetes, reduces blood sugar levels. This study will examine whether taking metformin with the antidepressant medication sertraline will enhance the effectiveness of sertraline in people who are overweight and depressed.

Participation in this study will last a total of 16 weeks and will include baseline testing and ten scheduled study visits. Participants will be randomly assigned to receive either sertraline and metformin or sertraline and placebo on a daily basis. The baseline visit will include the following tests and measures: an electrocardiogram (EKG), which will measure the electrical activity in the heart; an oral glucose tolerance test (OGTT), which will measure how a person's body breaks down glucose; a blood test, which will measure lipids, glycosylated hemoglobin (A1C), and other cardiometabolic risk factors; a dual energy x-ray absorptimetry (DEXA) scan, which will measure body fat; a pregnancy test for women; measurements of vital signs, height, weight, waist-to-hip ratio, and waist circumference; and questionnaires concerning health, medication use, physical activity, diet, and mood. Some of the questionnaires will be administered through interviews with a researcher. During the study visits, which will occur every 2 weeks, participants will complete questionnaires, unused medication will be collected, and new medication will be handed out. At Week 8, participants will provide an additional blood sample by finger stick.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than 28.7
* Positive screening for depression
* Must live within 100 miles of the St. Louis metropolitan area

Exclusion Criteria:

* Pregnant or breastfeeding
* Known hypersensitivity to sertraline or metformin
* Recent history of heart attack or unstable heart disease
* Severe liver disease or kidney impairment, defined by a serum creatine level above 3 mg/dL
* Psychiatric disorder thought to affect management, such as schizophrenia, or alcohol or drug dependence

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2007-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Lustman, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sertraline Plus Metformin: Participants will receive sertraline and metformin for 16 weeks.
  Sertraline: 50 mg once a day, which may be increased to 200 mg once a day
  Metformin: Starting dose of 500 mg daily and increasing by 500 mg every 2 weeks to a total of 2,000 mg daily
- Sertraline Plus Placebo: Participants will receive sertraline and placebo for 16 weeks.
  Sertraline: 50 mg once a day, which may be increased to 200 mg once a day
Period: Overall Study
Arm/Group | Sertraline Plus Metformin | Sertraline Plus Placebo
Started | 104 | 102
Completed | 66 | 62
Not Completed | 38 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline Plus Metformin | Sertraline Plus Placebo | Total
Number analyzed (Participants) | 104 | 102 | 206
Age, Continuous [Mean (Full Range); unit: years] | 43.67 [20 to 60] | 42.15 [22 to 58] | 42.91 [20 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 85 | 171
  Male | 18 | 17 | 35
Region of Enrollment [Number; unit: participants]
  United States | 104 | 102 | 206
Marital Status (married) [Number; unit: participants] | 48 | 45 | 93
Education [Mean (Full Range); unit: years] | 14.64 [10 to 18] | 14.60 [8 to 20] | 14.62 [8 to 20]
Baseline Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 38.53 [27.44 to 59.23] | 38.07 [27.80 to 58.42] | 38.30 [27.44 to 59.23]

OUTCOME MEASURES:

1. Primary Outcome: Change of Beck Depression Inventory-II Scores Over 16 Weeks
Description: Beck Depression Inventory-II (BDI) scores 0-63, minimum score =0, maximum score =63, Higher scores represent worse outcome. Baseline scores are compared to scores after treatment.
Time Frame: Measured at Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline Plus Metformin | Sertraline Plus Placebo
Number analyzed (Participants) | 104 | 102
units on a scale
  BDI Change Scores | 18.82 (8.78) | 17.50 (7.94)
  BDI at Baseline | 22.68 (8.00) | 22.03 (7.71)
  BDI at Week 16 | 3.86 (4.57) | 4.53 (4.10)
Statistical Analysis 1: Comparison: Sertraline Plus Metformin vs Sertraline Plus Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Sertraline Plus Metformin | Sertraline Plus Placebo
Serious Adverse Events (participants affected / at risk) | 0/104 | 1/102
Other Adverse Events (participants affected / at risk) | 44/104 | 41/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline Plus Metformin (N=104) | Sertraline Plus Placebo (N=102)
Syncopal episode leading to inpatient hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — Participant (pt) seen in ER- had a syncopal episode and fell at home. Later possible persecutory delusions & hyper-religiosity symptoms questioned; pt found walking "aimlessly" in traffic- transferred to psychiatric unit for admission and evaluation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sertraline Plus Metformin (N=104) | Sertraline Plus Placebo (N=102)
Headache (Nervous system disorders) | 28 | 32
Insomnia (Nervous system disorders) | 35 | 33
Fatigue (Nervous system disorders) | 42 | 36
Dizziness (Ear and labyrinth disorders) | 9 | 8
Weakness (General disorders) | 14 | 10
Diarrhea (Gastrointestinal disorders) | 28 | 22
Nausea (Gastrointestinal disorders) | 15 | 11
Flatulence (Gastrointestinal disorders) | 25 | 21
Indigestion (Gastrointestinal disorders) | 26 | 20
Bloating (Gastrointestinal disorders) | 24 | 14
Anorexia (Gastrointestinal disorders) | 7 | 8
Sexual Dysfunction (Vascular disorders) | 20 | 17
Sweating (Nervous system disorders) | 27 | 19
Tremors (Nervous system disorders) | 10 | 8
Dry mouth (General disorders) | 18 | 13
Constipation (Gastrointestinal disorders) | 8 | 12
Skin Itching (Skin and subcutaneous tissue disorders) | 16 | 10
Change in Hearing (Ear and labyrinth disorders) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No